CLINICAL TRIAL: NCT04455945
Title: Comparison of Quality of Life Outcomes Between Laparoscopic and Open Approach for Rectal Cancer Surgery
Brief Title: Quality of Life After Rectal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ramazan Sari, Principal Investigator, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: 2017/514/108/12
Record Dates: First submitted 2020-06-19; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Rectal Cancer; Quality of Life
Keywords: rectal cancer surgery; life quality; questionnaire
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open: Patients with open surgery for rectal cancer planned in our department.
  Interventions: Procedure: Open Rectal cancer surgery
- Laparoscopic: Patients with laparoscopic surgery for rectal cancer planned in our department.
  Interventions: Procedure: Laparoscopic Rectal cancer surgery

INTERVENTIONS:
Procedure: Open Rectal cancer surgery — Open sphincter preserving surgery for rectal cancer
  Groups: Open
Procedure: Laparoscopic Rectal cancer surgery — Laparoscopic sphincter preserving surgery for rectal cancer
  Groups: Laparoscopic

SUMMARY:
Following colorectal surgery, many patients face a combination of physical and emotional problems for a long period of time. Symptoms such as pain, fatigue, and disturbed bowel and sexual function, as well as problems in social and role functioning, inevitably affect the patients' well-being. Therefore, evaluation of the self-reported quality of life (QoL) is becoming increasingly important in clinical trials. The investigators aimed to compare long term health related life quality (HRQoL) results of laparoscopic approach with open approach in patients with sphincter preserving resections for rectal cancer at a single-center.

DETAILED DESCRIPTION:
This study is planned prospectively. All patients scheduled for operation due to rectal cancer in our clinic between January 2017 and December 2018 will be evaluated for suitability for the study. During the preoperative examination, patients will be informed about the study and their written consent will be obtained. Patients will be randomized between open and laparoscopic groups in the ratio 2:1, depending on the type of surgery. Clinical data of patients will be analyzed from the hospital database programme.

The EORTC QLQ-C30 and QLQ-CR29 questionnaires prepared by The European Organization for Research and Treatment of Cancer (EORTC) will be used to evaluate the quality of life after the operation. The EORTC QLQ-C30 questionnaire will be completed by examining the patients' daily observation notes. EORTC QLQ-CR29 will be completed with face to face interviews in the first year after surgery.

In this way, it will be aimed to compare the early and long-term quality of life (HRQoL) results of open and laparoscopic approach in patients undergoing surgery for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent surgery (laparoscopic or open) for rectal cancer in our department.

Exclusion Criteria:

* The patients whose all oncological treatments had not been completed at least 6 months ago
* The patients with ASA IV score
* The patients with previous abdominal surgery
* The patients who had developed major surgical complications (such as anastomosis leakage, requiring re-laparotomy, evisceration)
* The patients who underwent a new abdominal surgery except for stoma closure
* The patients with local recurrence or distant metastases
* The patients who still had a stoma
* The patients who did not want to take part in the study
* The patients who missed in the follow-up period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who underwent surgery (laparoscopic or open) for rectal cancer in our department.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Age | Before surgery
  Years
Gender | Before surgery
  Male/Female
BMI | Before surgery
  kg/m²
ASA | Before surgery
  I, II, III, IV
Tumor Localization | During the operation
  Upper/Middle/Low
Pathologic Stage | up to 10 days after surgery
  1A, 1B, 2A, 2B, 3A, 3B, 3C
Complications | Through study completion, an average of 1 year
  yes/no
European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire 30 (EORTC QLQ-C30) Functional scales | During one week after surgery
  Global/Physical/Role/Cognitive/Social functioning. All scales and single-item measurements range from 0 to 100. A higher score on a functional scale indicates better functioning.
European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire 30 (EORTC QLQ-C30) Symptom scales | During one week after surgery
  Fatigue/Nausea and vomiting/Pain/Dyspnoea/Insomnia/Appetite loss/Constipation/Diarrhoea/Financial difficulties. All scales and single-item measurements range from 0 to 100. A higher score for a symptom scale / item indicates a higher symptomatology and problem level.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Colorectal Cancer 29 (EORTC QLQ-CR29) Functional scales | During one year after surgery
  Body Image/Future projections/Weight/Sexual interest. All scales and single-item measurements range from 0 to 100. A higher score on a functional scale indicates better functioning.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Colorectal Cancer 29 (EORTC QLQ-CR29) Symptom scales | During one year after surgery
  Urinary frequency/Blood and mucus in stool/Stool frequency/Urinary incontinence/Dysuria/Abdominal pain/Buttock pain/Bloating/Dry mouth/Hair loss/Taste/Flatulence/Faecal incontinence/Sore skin/Embarrassment/Impotence/Dyspareunia. All scales and single-item measurements range from 0 to 100. A higher score for a symptom scale / item indicates a higher symptomatology and problem level.

CONTACTS AND LOCATIONS:
Overall Officials: Selcuk Kaya, MD, Study Chair — Kartal Dr. Lutfi Kirdar Training and Research Hospital
Locations (1):
- Kartal Dr Lutfi Kirdar Tranining and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson J, Angenete E, Gellerstedt M, Angeras U, Jess P, Rosenberg J, Furst A, Bonjer J, Haglind E. Health-related quality of life after laparoscopic and open surgery for rectal cancer in a randomized trial. Br J Surg. 2016 Nov;103(12):1746. doi: 10.1002/bjs.10280. Epub 2016 Jul 6. No abstract available. PMID 27801927
- [Background] D'Ambrosio G, Paganini AM, Balla A, Quaresima S, Ursi P, Bruzzone P, Picchetto A, Mattei FI, Lezoche E. Quality of life in non-early rectal cancer treated by neoadjuvant radio-chemotherapy and endoluminal loco-regional resection (ELRR) by transanal endoscopic microsurgery (TEM) versus laparoscopic total mesorectal excision. Surg Endosc. 2016 Feb;30(2):504-511. doi: 10.1007/s00464-015-4232-8. Epub 2015 Jun 5. PMID 26045097
- [Background] D'Ambrosio G, Picchetto A, Campo S, Palma R, Panetta C, De Laurentis F, La Rocca S, Lezoche E. Quality of life in patients with loco-regional rectal cancer after ELRR by TEM versus VLS TME after nChRT: long-term results. Surg Endosc. 2019 Mar;33(3):941-948. doi: 10.1007/s00464-018-6583-4. Epub 2018 Nov 12. PMID 30421081